CLINICAL TRIAL: NCT00912795
Title: SMS Turkey: Harnessing the Power of TXT Messaging to Promote Smoking Cessation
Brief Title: SMS Turkey: Harnessing the Power of Text Messaging to Promote Smoking Cessation
Acronym: SMS Turkey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Innovative Public Health Research (Other)
Collaborators: Hacettepe University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ISK-NIH-FIC7918; 5R01TW007918 (NIH)
Record Dates: First submitted 2009-05-19; First posted 2009-06-03 (Estimated); Results first posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-08

CONDITIONS: Smoking
Keywords: Smoking Cessation; technology; developing countries
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS Turkey (Experimental): 6-week smoking cessation program delivered via daily text messages
  Interventions: Behavioral: SMS Turkey
- Brochure control (No Intervention): 7-page brochure that provided general information and tips on how to quit smoking

INTERVENTIONS:
Behavioral: SMS Turkey — 6-week smoking cessation program delivered via daily text messages
  SMS Turkey: 6-week smoking cessation program delivered via text messaging. SMS Turkey content is guided by the Cognitive Behavioral Therapy (CBT) theory.
  Content was tailored based on participant's stage in quitting (i.e., pre-quit, quit day, early-quit, late-quit, relapse). Based on the typical relapse trajectory, content paths were created for participants based on whether or not they were smoking 2 days after quit day; and again at 7 days after quit day.
  Depending on the participant's content path, the total number of messages received ranged from 91 (for those assigned to the encouragement arm) to 146 (for those who relapsed and then were assigned to the late quit messages).
  Other Names: Cebiniz birakin diyor
  Arms: SMS Turkey

SUMMARY:
The purpose of this study is to develop and test a text messaging-based smoking cessation program for adults who are currently smoking and want to quit, living in Turkey.

DETAILED DESCRIPTION:
Smoking has long been recognized as a significant public health concern associated with great morbidity and mortality. Although smoking rates have decreased in high income countries, these trends have not been noted for tow and middle income countries. This is especially true in Turkey, which was ranked 6th in the world in smoking consumption. Between 51-63% of Turkish men and 24-26% of Turkish women 15 years of age and older are smokers. With lung cancer the leading cancer-related cause of death for both men and women, effective and accessible smoking cessation interventions are needed. Cell phone technology represents a unique opportunity to deliver evidenced-based smoking cessation behavioral treatments through a delivery mechanism already widely adopted by adults. An estimated 35 million Turks were using cell phones, making them 1.8 times more common than land lines. Cell phone interventions are a unique delivery method because of their 'always on' capability. The rapid uptake of cell phones allows us to potentially reach those who might otherwise not utilize smoking cessation services.

We designed and evaluated SMS Turkey, an evidenced-based smoking intervention that takes advantage of technologies adopted by adult smokers in Turkey. The primary outcome measure is sustained abstinence 12 weeks after quit day, confirmed with a carbon monoxide (CO) reading of 8 ppm or less. Sustained abstinence was defined as 5 or fewer cigarettes smoked since the quit date, per West et al. Secondary outcome measures included: 7-day and 30-day point prevalence of smoking behavior at 3 months; CO-verified 7-day point prevalence at 4 weeks; and reduction in cigarettes per day for those who are smoking at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently smoking every day
* Owning a TXT-capable cell phone
* Sent or received TXT messages at least once in the past year
* Living in Ankara (to ease technology support if necessary)
* Agreement to set quit day in 15 days from enrollment date
* Agreement to verification of smoking cessation using a carbon monoxide breath monitor

Exclusion Criteria:

• No chronic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Ybarra, MPH PhD, Principal Investigator — Center for Innovative Public Health Research
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ybarra ML, Bagci Bosi AT, Bilir N, Holtrop JS, Korchmaros J, Emri S. Interest in technology-based and traditional smoking cessation programs among adult smokers in Ankara, Turkey. Tob Induc Dis. 2011 Aug 1;9(1):10. doi: 10.1186/1617-9625-9-10. PMID 21806793
- [Background] Ybarra ML, Holtrop JS, Bagci Bosi AT, Emri S. Design considerations in developing a text messaging program aimed at smoking cessation. J Med Internet Res. 2012 Jul 24;14(4):e103. doi: 10.2196/jmir.2061. PMID 22832182
- [Result] Ybarra M, Bagci Bosi AT, Korchmaros J, Emri S. A text messaging-based smoking cessation program for adult smokers: randomized controlled trial. J Med Internet Res. 2012 Dec 27;14(6):e172. doi: 10.2196/jmir.2231. PMID 23271159
- [Result] Ybarra ML, Holtrop JS, Bagci Bosi AT, Bilir N, Korchmaros JD, Salih Emri AK. Feasibility and acceptability of a text messaging-based smoking cessation program in ankara, Turkey. J Health Commun. 2013 Aug;18(8):960-73. doi: 10.1080/10810730.2012.757399. Epub 2013 Apr 29. PMID 23627304

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Ankara, Turkey between December 2010 & June 2011, through in-person outreach at local shopping malls and local newspapers advertisements. Flyers were also posted at Hacettepe University. Smokers indicated their interest by calling the study office or speaking directly with the research assistant at the shopping mall.
Pre-assignment Details: Of the 247 people who expressed interest in participating, 230 were eligible for the study. A total of 151 adults (66% of those eligible) attended the enrollment meeting, where they consented to take part in the research study and were randomly assigned to either the intervention or control group.
Groups:
- Brochure Control: A 7-page brochure that provided general information and tips on how to quit smoking. Participants did not receive any text messages.
  The brochure encouraged smokers to follow 5 steps to quitting : (1) set a quit day and sign a contract, (2) find out about their smoking patterns-why they smoke, (3) practice quitting and change their patterns, (4) involve their family and friends, and (5) learn to be a self-supporter.
Period: Overall Study
Arm/Group | SMS Turkey | Brochure Control
Started | 76 | 75
Completed | 29 | 17
Not Completed | 47 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMS Turkey | Brochure Control | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.3) | 36.1 (9.5) | 35.89 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 24 | 59
  Male | 41 | 51 | 92
Income [Number; unit: participants]
  Less than 2000 Turkish lira per month | 23 | 37 | 60
  2000 - 4000 Turkish lira per month | 34 | 28 | 62
  More than 4000 Turkish lira per month | 16 | 9 | 25
  Do not want to answer | 3 | 1 | 4
Martial status [Number; unit: participants]
  Married | 42 | 49 | 91
  Single | 30 | 25 | 55
  Divorced | 4 | 0 | 4
  Widowed | 0 | 1 | 1
Educational attainment [Number; unit: participants]
  High school or less | 28 | 38 | 66
  Two-year college | 13 | 10 | 23
  University degree | 27 | 23 | 50
  Post graduate degree | 8 | 4 | 12
Average Number of cigarettes smoked per day [Mean (Standard Deviation); unit: number of cigarettes per day] | 18.7 (7.2) | 20.4 (9.2) | 19.53 (8.27)
Age at first cigarette [Mean (Standard Deviation); unit: years] | 17.5 (3.7) | 17.1 (3.6) | 17.3 (3.6)
Fagerström score [Mean (Standard Deviation); unit: score] — Tobacco dependence was assessed using the Fagerström Test of Nicotine Dependence (FTND). Scores range from 0-10. A score of 0-2 indicates low dependence, 3-4 indicates low to moderate dependence, 5-7 indicates moderate dependence, and 8-10 indicates high dependence.
  score | 4.8 (2.3) | 4.9 (2.5) | 4.8 (2.4)
Importance of quitting to self [Mean (Standard Deviation); unit: score] — This measure has scores possibly ranging form 4 to 10 with higher scores reflecting more importance
  score | 8.9 (1.6) | 9.0 (1.4) | 8.9 (1.5)
Confidence in one's ability to quit [Mean (Standard Deviation); unit: score] — This measure has scores possibly ranging form 0 to 10 with higher scores reflecting more confidence
  score | 6.0 (2.4) | 6.0 (2.5) | 6.0 (2.5)
Number of quit attempts in the past year [Mean (Standard Deviation); unit: number of quit attempts] | 2.4 (1.5) | 2.4 (1.5) | 2.4 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Carbon Monoxide-verified Continuous Abstinence at 12 Weeks
Description: self-reported continuous abstinence since quit day (<=5 cigarettes) verified with carbon monoxide reading (<=8ppm)
Time Frame: 12-weeks post-quit day
Population: Intention-to-treat (ITT) analysis: All participants randomized at baseline included in analyses regardless of completion of 12-week follow-up data. Missing equals failure (i.e., smoked cigarettes).
Measure: Number; unit: participants
Arm/Group | SMS Turkey | Brochure Control
Number analyzed (Participants) | 76 | 75
participants | 8 | 4
Statistical Analysis 1: Comparison: SMS Turkey vs Brochure Control; Test type: Superiority or Other; Risk Ratio (RR) = 2.0, 95% CI 2-sided [0.62 to 6.3]

2. Secondary Outcome: CO-verified 7-day Point Prevalence Abstinence at 4 Weeks
Description: self-reported continuous abstinence in the past 7 days at 4 weeks (<=5 cigarettes) verified with carbon monoxide reading (<=8ppm)
Time Frame: 4 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SMS Turkey | Brochure Control
Number analyzed (Participants) | 76 | 75
participants | 9 | 7
Statistical Analysis 1: Comparison: SMS Turkey vs Brochure Control; Test type: Superiority or Other; Risk Ratio (RR) = 1.3, 95% CI 2-sided [0.50 to 3.2]

3. Secondary Outcome: Self-reported 7-day Point Prevalence Abstinence at 12 Weeks
Description: self-reported smoking abstinence in the past 7 days at 12 weeks (<=5 cigarettes)
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SMS Turkey | Brochure Control
Number analyzed (Participants) | 76 | 75
participants | 10 | 4
Statistical Analysis 1: Comparison: SMS Turkey vs Brochure Control; Test type: Superiority or Other; Risk Ratio (RR) = 2.5, 95% CI 2-sided [0.81 to 7.5]

4. Secondary Outcome: Self-reported 30-day Point Prevalence Abstinence at 12 Weeks
Description: self-reported smoking abstinence in the past 30 days at 12 weeks (<=5 cigarettes)
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | SMS Turkey | Brochure Control
Number analyzed (Participants) | 76 | 75
participants | 8 | 4
Statistical Analysis 1: Comparison: SMS Turkey vs Brochure Control; Test type: Superiority or Other; Risk Ratio (RR) = 2.0, 95% CI 2-sided [.62 to 6.3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through the study period (i.e., from baseline to 12-week follow-up).
Arm/Group | SMS Turkey | Brochure Control
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75

LIMITATIONS AND CAVEATS:
An imbalance favoring the intervention was detected after approximately 100 participants were enrolled. To ensure a 1:1 match, the procedure was modified so that the RA pulled a slip of paper from a hat that read either "SMS Turkey" or "brochure."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No